CLINICAL TRIAL: NCT05624762
Title: The Therapeutic Effect of Low-intensity Focused Ultrasound on Painful Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qian Ge, Professor, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPN-China2022
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Painful Diabetic Neuropathy; low-intensity focused ultrasound
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIFU group (Active Comparator): receive LIFU therapy
  Interventions: Device: Low-Intensity Focused Ultrasound (LIFU)
- Control group (Sham Comparator): receive sham LIFU therapy
  Interventions: Device: Sham Low-Intensity Focused Ultrasound

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound (LIFU) — LIFU device (LCA200; Chongqing Haifu Medical Technology Co., Ltd., Chongqing, China).
  Arms: LIFU group
Device: Sham Low-Intensity Focused Ultrasound — Sham Low-Intensity Focused Ultrasound
  Arms: Control group

SUMMARY:
Diabetic painful peripheral neuropathy (DPN) constitutes a serious threat to the outcomes of patients with diabetes. Yet, the treatments for targeting the underlying nerve damage and relieving pain are limited. The low-intensity focused ultrasound (LIFU) has been demonstrated to regulate neuronal activity without any concomitant tissue damage. Studies in animal models have shown that LIFU could protect nerve cells against inflammation and oxidative stress, as well as stimulate neurotrophic factor production. In humans, LIFU has been reported to be effective in relieving peripheral neurogenic pain caused by carpal tunnel syndrome and chemotherapy drugs. Thus, we aim to design a randomized controlled double-blind study by using LIFU. The primary endpoint is the patient's pain score (NRS), and the secondary endpoints include Neuropathy Symptom Score (NSS) and Neuropathy Deficit Score (NDS). Through this study, we anticipate establishing a new method for managing painful DPN.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) is a major cause of disability and mortality due to pain, loss of protective sensation, foot ulceration, amputation, and risk of falls, therefore constituting a serious threat to the outcomes of patients with diabetes and their treatment costs. The pathogenesis of DPN has been proposed as an inflammatory and oxidative stress injury in nerve cells caused by glucose and lipid metabolism disorder. Yet, the treatments for targeting the underlying nerve damage and relieving pain are limited. The widely used drugs such as Mecobalamine and Lipoic acid are not effective in some patients (about 2/3). Others, like anticonvulsant (e.g. Dabapentin), antidepressant (e.g. Duloxetine), and central opioid analgesics (e.g. Tramadol), are effective in the short-term, but they may lead to side effects for long-term use such as impairment of cognitive function, insomnia, and addiction, etc. The low-intensity focused ultrasound (LIFU) is regarded as the magnitude of ultrasonic intensity similar to or below that typically used in diagnostic ultrasound examinations. Although currently LIFU has not been applied in DPN, a number of studies have demonstrated that it can regulate neuronal activity without any concomitant tissue damage. Studies in animal models have shown that LIFU could protect nerve cells against inflammation and oxidative stress, as well as stimulate neurotrophic factor production. In humans, LIFU has been reported to be effective in relieving pain caused by carpal tunnel syndrome (Median nerve compression). Also, several studies have evidenced that cancer patients suffering from chemotherapy drug-induced peripheral neurogenic pain had significant improvement by LIFU treatment. Thus, we aim to take advantage of LIFU to treat the painful DPN. We plan to design a randomized controlled double-blind study. The primary endpoint is the patient's pain score (NRS), and the secondary endpoints include Neuropathy Symptom Score (NSS) and Neuropathy Deficit Score (NDS). Through this study, we anticipate establishing a new method for managing painful DPN.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 80 years
* having diabetes based on the criteria of the World Health Organization (WHO 1999)
* Having diabetic painful neuropathy for more than 1 month but less than 5 years
* no alcohol addiction (consumption<140g/week in men and <70g/week in women)
* no history of cerebral infarction/hemorrhage or other known nervous system disease
* no active infections in the skin

Exclusion Criteria:

* having abnormalities in levels of Vitamin B12, Hemoglobin, and TSH.
* HbA1C>10%
* having moderate or severe hepatic and renal dysfunctions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
pain score | 7 days
  the pain score is evaluated using a numeric pain rating (0-10) scale (NRS)

SECONDARY OUTCOMES:
Neuropathy Symptom Score (NSS) | 7 days
  the NSS is determined using a questionnaire
Neuropathy Deficit Score (NDS) | 7 days
  the NDS is examined by an experienced neurologist

OTHER OUTCOMES:
The motor nerve conduction velocity (MNCS) | 7 days
  The motor nerve conduction velocity (MNCS) measured in peroneal, tibial, and sural nerves using electromyography
The sensory nerve conduction velocity (SNCS) | 7 days
  The sensory nerve conduction velocity (SNCS) were measured in peroneal, tibial, and sural nerves using electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Qian Ge, Professor, Study Director — Department of Endocrinology, the First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No